CLINICAL TRIAL: NCT05576519
Title: Immunohistochemical Expression of Epithelial Cell Adhesion Molecule (EpCAM) in Epithelial Ovarian Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Abd El-Sadek Ahmed, Lecturer at Pathology Department, Faculty of Medicine, Sohag University
Other Study IDs: Soh-Med-22-09-15
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Carcinoma
Keywords: Ovarian carcinoma; CSCs; EpCAM
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer stem cells (CSCs) can undergo self-renewal and differentiation. EpCAM is a 40-kDa type I transmembrane glycoprotein composed of a large extracellular domain, one transmembrane region, and a small intracellular domain of 26 amino acids. Recent insights revealed that it is involved in promoting cancer cell proliferation, migration, and invasiveness. It is used as a diagnostic and prognostic marker. EpCAM has also recently been identified as a marker for CSCs.

DETAILED DESCRIPTION:
Ovarian carcinoma is one of most frequent cancer in women worldwide. Epithelial ovarian carcinoma is a group of neoplasms with different histologic pictures. Serous carcinoma is the most common type.

Cancer stem cells (CSCs) can undergo self-renewal and differentiation. EpCAM is a 40-kDa type I transmembrane glycoprotein composed of a large extracellular domain, one transmembrane region, and a small intracellular domain of 26 amino acids. It is abundantly expressed by the majority of human epithelial carcinomas, including colorectal, breast, lung, prostate, ovarian, and endometrial cancers. it is overexpressed in various neoplasms. Recent insights revealed that it is involved in promoting cancer cell proliferation, migration, and invasiveness. It is used as a diagnostic and prognostic marker. EpCAM has also recently been identified as a marker for CSCs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epithelial ovarian carcinoma and underwent surgery

Exclusion Criteria:

* - Cases received pre-operative chemotherapy or radiotherapy.
* Cases with insufficient clinical data.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Fifty paraffin blocks of EOC collected from the archive of Pathology Department of Sohag Faculty of Medicine during the time period from June 2017 to June 2022.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
evaluate EpCAM expression in ovarian carcinoma | 1 month
  IHC

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Sohag University, Sohag
  - Faculty of Medicine, Sohag